CLINICAL TRIAL: NCT05957263
Title: The Combined Effect of Biofeedback Training and Osteopathic Procedures for the Treatment of Functional Daytime Urinary Incontinence: a Prospective, Randomized Clinical Trial
Brief Title: Biofeedback and Osteopathic Procedures for Daytime Urinary Incontinence
Acronym: BOFDUI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F.P.T 2307001
Record Dates: First submitted 2023-07-07; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Urinary Incontinence
Keywords: Biofeedback training; Osteopathic procedures; 24-hour pad test; functional daytime urinary incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: controlled, double-blinded, and randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: both participants and assessors will be blind for the treatment procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Biofeedback training and Osteopathy procedure (Experimental): the biofeedback training lasts 10 weeks and involves 3 sessions per week, with each session lasting for 15 minutes. During biofeedback-assisted pelvic floor muscle exercises, the child was asked to contract the pelvic floor muscles as if stopping peeing, after which the biofeedback device helps them understand how to better control their muscles.
  The osteopathy techniques involved a combination of myofascial, visceral, and articular techniques aimed at restoring and rebalancing internal tensions and improving visceral mobility.
  Interventions: Other: Biofeedback training and Osteopathy procedure; Other: Biofeedback training; Other: Osteopathy procedure
- Biofeedback training (Active Comparator): he biofeedback training lasts 10 weeks and involves 3 sessions per week, with each session lasting for 15 minutes. During biofeedback-assisted pelvic floor muscle exercises, the child was asked to contract the pelvic floor muscles as if stopping peeing, after which the biofeedback device helps them understand how to better control their muscles.
  Interventions: Other: Biofeedback training
- Osteopathy procedure (Active Comparator): The osteopathy techniques involved a combination of myofascial, visceral, and articular techniques aimed at restoring and rebalancing internal tensions and improving visceral mobility.
  Interventions: Other: Osteopathy procedure

INTERVENTIONS:
Other: Biofeedback training and Osteopathy procedure — the biofeedback training lasts 10 weeks and involves 3 sessions per week, with each session lasting for 15 minutes. the child was asked to contract the pelvic floor muscles as if stopping peeing, after which the biofeedback device helps them understand how to better control their muscle. muscle inhibition for the psoas muscle, deep massages in the obturator foramen, stretching for the greater omentum, and abdominal maneuvers. a high velocity, low amplitude manipulation performed for the sacroiliac joint and T10-L2 region. The treatments were implemented in phases, with multiple sessions for each phase over a 10-week period. Each osteopathy session typically lasted 30 minutes, with the myofascial, visceral, and articular techniques performed twice a week for 15 minutes each session for 10 weeks, and the high velocity, l
  Other Names: BTOP
  Arms: Biofeedback training and Osteopathy procedure
Other: Biofeedback training — the biofeedback training lasts 10 weeks and involves 3 sessions per week, with each session lasting for 15 minutes. During biofeedback-assisted pelvic floor muscle exercises, the child was asked to contract the pelvic floor muscles as if stopping peeing, after which the biofeedback device helps them understand how to better control their muscles.
  Other Names: BIOFB
  Arms: Biofeedback training; Biofeedback training and Osteopathy procedure
Other: Osteopathy procedure — specific techniques included muscle inhibition for the psoas muscle, deep massages in the obturator foramen, stretching for the greater omentum, and abdominal maneuvers. In addition, there was a high velocity, low amplitude manipulation performed for the sacroiliac joint and T10-L2 region. The treatments were implemented in phases, with multiple sessions for each phase over a 10-week period. Each osteopathy session typically lasted 30 minutes, with the myofascial, visceral, and articular techniques performed twice a week for 15 minutes each session for 10 weeks, and the high velocity, low amplitude manipulation performed three times a week for 15 minutes each session for 10 weeks.
  Other Names: OSP
  Arms: Biofeedback training and Osteopathy procedure; Osteopathy procedure

SUMMARY:
The study will enroll 113 participants, randomly will be assigned to one of three groups will receive either group A will receive combined therapy of biofeedback training and osteopathy techniques, group B will receive biofeedback training, group C will receive osteopathy technique only over a period of 10 weeks, followed by an 8-week follow-up period. Outcome measures will include the 24-hour pad test, Pediatric Lower Urinary Tract Symptom Score (PLUTSS), and the bladder diary.

DETAILED DESCRIPTION:
Children (male and female) with functional daytime urinary incontinence, typically the urge type, who were referred for physical therapy by a urologist were recruited from Mansoura Urology and Nephrology Hospital at Mansoura University. To participate in the study, participants had to be between 6 and 16 years old and have had functional daytime urinary incontinence for at least six months, with at least three episodes per week and a total of at least 60 ml of urine loss per week. Certain exclusion criteria were applied, including not having other types of urinary incontinence, neurological disorders, previous operations on the urinary or bowel system, current use of certain medications that could interfere with study results or pose a risk to the participant's health, severe cognitive impairment or dementia, recent participation in another clinical trial, active urinary tract infection (UTI), not having vascular disorders in the urinary system, and parental refusal to sign the written consent form.

ELIGIBILITY:
Inclusion Criteria:

* between 6 and 16 years old
* have functional daytime urinary incontinence for at least six months
* at least three episodes per week

Exclusion Criteria:

* neurological disorders,
* previous operations on the urinary or bowel system
* current use of certain medications that could interfere with study results
* pose a risk to the participant's health
* severe cognitive impairment or dementia

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 117 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
The 24-hour pad test | 10 weeks
  The pad is weighed at the beginning and end of the test to determine the amount of urine leakage, which is used to estimate the severity of the condition and evaluate the effectiveness of the treatment. Several studies have been used to assess the test-retest reliability of the 24-hour pad test and found it to be a reliable tool for the diagnosis and monitoring of urinary incontinence

SECONDARY OUTCOMES:
Pediatric Lower Urinary Tract Symptom Score | 10 weeks
  The PLUTSS is a questionnaire used to evaluate lower urinary tract symptoms (LUTS) in children by assessing the frequency and severity of urinary symptoms including urgency, frequency, incontinence, and urinary tract infections. Both children and their parents provide responses, and the scoring ranges from 0-34, with higher scores indicating more severe symptoms. A score of 0-5 is normal, 6-10 is mild, 11-20 is moderate, and 21-34 indicates severe symptoms
Assessment of the frequency of daytime urinary incontinence | 10 weeks
  Monitoring the frequency of daytime urinary incontinence typically involves maintaining a bladder diary, which is a log of the patient's urination patterns indicating the number of times urination occurs, the amount of urine voided, and the presence of urinary incontinence episodes throughout the day.

CONTACTS AND LOCATIONS:
Locations (1):
- Hany Mohamed Elgohary, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
i have no intent to share my results

REFERENCES:
- [Result] Elgohary HM, Al Jaouni SK, Selim SA. Effect of ultrasound-enhanced Nigella sativa seeds oil on wound healing: An animal model. J Taibah Univ Med Sci. 2018 Jun 27;13(5):438-443. doi: 10.1016/j.jtumed.2018.02.008. eCollection 2018 Oct. PMID 31435359